CLINICAL TRIAL: NCT02944578
Title: Biomolecular Effects of Topical Curcumin in HSIL Cervical Neoplasia
Brief Title: Topical Curcumin for Precancer Cervical Lesions
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to patient feedback and need to redesign the delivery method.
Sponsor: Lisa Flowers (Other)
Responsible Party: Sponsor-Investigator, Lisa Flowers, Professor, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00079183
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Neoplasms
Keywords: Cancer; HIV; Oncology; Infectious Diseases; HPV; Preventive Medicine
MeSH Terms: conditions — Neoplasms; Communicable Diseases | interventions — Curcumin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Curcumin Arm (Experimental): Participants in this arm will use 2000 mg of intravaginal curcumin once a week for 12 weeks.
  Interventions: Drug: Curcumin
- Placebo Arm (Placebo Comparator): Participants in this arm will use 2000 mg of a placebo once a week for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Curcumin — Curcumin (Curcumin C3 Complex®, prepared by Sabinsa Corporation), a constituent of the spice turmeric, is considered to be a low-toxicity, dietary-derived agent with chemopreventive and therapeutic benefits.
  Study participants will be instructed to insert four 500 mg (2000 mg total) curcumin capsules once a week (excluding days when they are on their menses). Participants will insert the capsules using the vaginal applicator while lying on their back with their knees bent. Participants will be instructed to gently insert the capsules into the vagina as far as they will go comfortably, similar to a tampon insertion or other common intravaginal drugs.
  Cervical cytology, colposcopies and biopsies will be performed at the Baseline, Week 4, 8, 12 and 16 visits to collect samples to analyze for the study outcomes.
  Other Names: Curcumin C3 Complex
  Arms: Curcumin Arm
Drug: Placebo — Study participants randomized to the placebo arm will insert four 500 mg (2000 mg total) of the placebo (gelatin) capsules once a week (excluding days when they are on their menses). Participants will insert the capsules using the vaginal applicator while lying on their back with their knees bent. Participants will be instructed to gently insert the capsules into the vagina as far as they will go comfortably, similar to a tampon insertion or other common intravaginal drugs.
  Cervical cytology, colposcopies and biopsies will be performed at the Baseline, Week 4, 8, 12 and 16 visits to collect samples to analyze for the study outcomes.
  Arms: Placebo Arm

SUMMARY:
The purpose of this study is to see if curcumin can reverse a cervical precancerous state by looking at people who have the condition and intervening with a study drug or placebo (an inactive drug), prior to planned therapeutic loop electrosurgical excision procedure (LEEP) which is a treatment procedure for removing cervical cancer. 40 women with high grade squamous intraepithelial lesion (HSIL) of the cervix will be enrolled to either insert 2000 mg capsule of curcumin or a placebo in their vagina once a week for 12 weeks. After a 4 week long washout period the participants will then undergo removal of the precancerous cells as recommended standard of care. Participants will have regular monthly visits for the duration of the study.

DETAILED DESCRIPTION:
Cervical cancer is the third most common cancer worldwide. The causative agent responsible for cervical cancer is the persistent infection with oncogenic Human Papillomavirus (HPV). Rates of cervical cancer and HPV infection are increased in HIV-infected women due to immunosuppression and cervical cancer is an AIDS-defining diagnosis. Despite the promise of HPV vaccine in the prevention of cervical cancer, the widespread availability of this vaccine is limited due to cost and accessibility. Therefore, prevention strategies to reduce cervical cancer after HPV exposure entail treatment at the most severe premalignant state (high grade squamous intraepithelial lesion or HSIL). As this procedure is expensive and not widely available in resource-limited areas there is a need for an inexpensive, non-invasive alternative method to treat these premalignant cervical lesions.

Curcumin, an extract from turmeric, a popular culinary spice, has been used in traditional Indian medicine for its anti-inflammatory and anti-infectious properties. Recent studies have shown the potential effect of curcumin to reduce tumors and precancerous lesions in animal and human cancer cells. It is postulated that curcumin achieves its effect on cancer cells by modulating different cellular pathways as well as altering HPV effect on tissue cells.

This study will explore the effect of curcumin as a potential medical treatment in HIV-infected women with HSIL lesions of the cervix. 40 women with high grade squamous intraepithelial lesion (HSIL) of the cervix will be enrolled to either insert 2000 mg capsule of curcumin or a placebo in their vagina once a week for 12 weeks. After a 4 week long washout period the participants will then undergo removal of the precancerous cells as recommended standard of care. Participants will have regular monthly visits for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive women and HIV negative women
* HSIL cytology with no invasive features identified on colposcopy or the baseline biopsy
* Compliant on combined antiretrovirals (cART)
* On continuous antiretrovirals with cluster of differentiation 4 (CD4) count >200 cells/ml with sustained undetectable viral load for at least 3 months
* Patient on reliable birth control. Adequate birth control includes: Combined oral contraceptive pill (OCP), Long Lasting Reversible Contraceptive (LARCP), BiLateral Tubal Ligation (BLT) and DepoProvera Shot/Birth control shot.
* Patient willing to conform to the study requirements
* No risk factors for microinvasive disease (no colposcopic features of microinvasion, adequate colposcopy and negative endocervical curettage)

Exclusion Criteria:

* Lactating and pregnant women
* Patient with irregular cycles (more than once a month).
* Previous hysterectomy and/or prior treatment for cervical precancer condition

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Flowers, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Grady Hospital - Ponce De Leon Clinic, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Grady Hospital Ponce De Leon Center in Atlanta Georgia, USA. Participant enrollment began November 20, 2017 and all follow-up assessments were completed by October 30, 2018. The study was suspended for several years due to participant feedback about using the suppository tablets and then the coronavirus disease 2019 (COVID-19) pandemic, and the study was ultimately terminated in April 2024.
Groups:
- Curcumin: Participants using 2000 mg of intravaginal curcumin capsules once a week for 12 weeks.
- Placebo: Participants using 2000 mg of intravaginal placebo capsules once a week for 12 weeks.
Period: Overall Study
Arm/Group | Curcumin | Placebo
Started | 4 | 3
Completed | 3 | 3
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Curcumin | Placebo | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Human Papillomavirus (HPV) Related Molecular Target HPV E6/E7 Messenger Ribonucleic Acid (mRNA) Expression Within HSIL Lesions of the Cervix
Description: Vaginal samples were used to determine the association between intravaginal curcumin on known HPV-related molecular target HPV E6/E7 mRNA expression within high grade squamous intraepithelial (HSIL) lesions of the cervix in HIV- infected women. The Aptima® HPV Assay that will be utilized detects full-length HPV E6/E7 mRNA for HPV types 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, and 68 and correlates very well with integrated HPV, which in turn correlates with full-length HPV E6/E7 protein levels.
Time Frame: Baseline, Weeks 4, 8, 12, and 16
Population: This analysis includes participants who attended the indicated study visit; some participants missed some visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 4 | 3
Participants
  Baseline | 0 | 1
  Week 4: number analyzed (Participants) | 2 | 3
  Week 4 | 0 | 0
  Week 8: number analyzed (Participants) | 2 | 3
  Week 8 | 0 | 0
  Week 12: number analyzed (Participants) | 3 | 2
  Week 12 | 0 | 0
  Week 16: number analyzed (Participants) | 2 | 3
  Week 16 | 0 | 0

2. Secondary Outcome: Curcumin Levels in Cervical Tissue
Description: Vaginal sampling and colposcopy with targeted cervical biopsies will be examined to establish the level of curcumin penetration in cervical tissue, as well as the cumulative effect of daily curcumin over time.
Time Frame: Weeks 4, 8, 12, and 16
Population: Study enrollment stopped early and the focus of the study shifted to analysis of the primary outcome measure among current participants. Samples for analysis of curcumin in cervical tissue were not collected from any participants.
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Explore the Association Between Curcumin and Nuclear Factor Kappa-light-chain-enhancer of Activated B Cells (NF-κB)
Description: Vaginal samples and cervical biopsies, obtained at each study visit, will be used to determine the association between curcumin and known biomarkers of cervical disease. This exploratory aim seeks to use repeated-measures analyses, utilizing a linear mixed model for the curcumin group to assess the association between nuclear factor kappa-light-chain-enhancer of activated B cells (NF-κB) and the concentration of curcumin at each time point. NF-κB upregulation is related to the grade of cervical intraepithelial neoplasia (CIN) although the significance of NF-κB activation per se to CIN lesion development and its prognostic value in cervical cancer have not been well defined. The analysis of NF-κB binding activity will provide a direct molecular benchmark for assessing curcumin treatment responses independent from its therapeutic effects.
Time Frame: Baseline, Weeks 4, 8, 12, and 16
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Explore the Association Between Curcumin and p16INK4a
Description: Vaginal samples and cervical biopsies, obtained at each study visit, will be used to determine the association between curcumin and known biomarkers of cervical disease. This exploratory aim seeks to use repeated-measures analyses, utilizing a linear mixed model for the curcumin group to assess the association between p16INK4a and the concentration of curcumin at each time point. p16INK4a (a tumor suppressor protein) is an indirect marker of cell cycle dysregulation and has been shown to be expressed in cervical dysplasias and carcinomas associated with high risk HPV infections.
Time Frame: Baseline, Weeks 4, 8, 12, and 16
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Explore the Association Between Curcumin and Rb
Description: Vaginal samples and cervical biopsies, obtained at each study visit, will be used to determine the association between curcumin and known biomarkers of cervical disease. This exploratory aim seeks to use repeated-measures analyses, utilizing a linear mixed model for the curcumin group to assess the association between Rb and the concentration of curcumin at each time point. Rb is an important cell cycle regulator protein in cervical carcinogenesis which is suppressed in most cervical cancer cells. Increased levels of this protein has been linked to regression of cervical cancer lesions.
Time Frame: Baseline, Weeks 4, 8, 12, and 16
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Explore the Association Between Curcumin and p53
Description: Vaginal samples and cervical biopsies, obtained at each study visit, will be used to determine the association between curcumin and known biomarkers of cervical disease. This exploratory aim seeks to use repeated-measures analyses, utilizing a linear mixed model for the curcumin group to assess the association between p53 and the concentration of curcumin at each time point. p53 is an important cell cycle regulator protein in cervical carcinogenesis which is suppressed in most cervical cancer cells. Increased levels of this protein have been linked to regression of cervical cancer lesions.
Time Frame: Baseline, Weeks 4, 8, 12, and 16
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Explore the Association Between Curcumin and Vascular Endothelial Growth Factor (VEGF)
Description: Vaginal samples and cervical biopsies, obtained at each study visit, will be used to determine the association between curcumin and known biomarkers of cervical disease. This exploratory aim seeks to use repeated-measures analyses, utilizing a linear mixed model for the curcumin group to assess the association between vascular endothelial growth factor (VEGF) and the concentration of curcumin at each time point. VEGF expression has been shown to correlate with severity of cervical intraepithelial neoplasia (CIN) lesions and invasive disease.
Time Frame: Baseline, Weeks 4, 8, 12, and 16
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time that participants gave consent to participant in the study continued through the final assessment at Week 16.
Arm/Group | Curcumin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-27): https://cdn.clinicaltrials.gov/large-docs/78/NCT02944578/Prot_SAP_000.pdf